CLINICAL TRIAL: NCT07066579
Title: Evaluation of the Effect of the Valsalva Maneuver on Invasive Pain During Arteriovenous Fistula Cannulation in Hemodialysis Patients
Brief Title: Evaluating the Effect of the Valsalva Maneuver on Invasive Pain During Arteriovenous Fistula Cannulation in Hemodialysis Patients
Acronym: VALPAIN-HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cansu POLAT DÜNYA (Other)
Collaborators: Istanbul University Scientific Research Projects Coordination Unit- Pending (Unknown)
Responsible Party: Sponsor-Investigator, Cansu POLAT DÜNYA, PhD, Associate Professor, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12.06.2025/3354894; 42077 (Other Grant/Funding Number: Istanbul University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Arteriovenous Fistula; Pain; Hemodialysis Access Failure; Vascular Access Device Complications
Keywords: Hemodialysis; Arteriovenous Fistula; Cannulation Pain; Valsalva Maneuver
MeSH Terms: conditions — Arteriovenous Fistula; Pain | interventions — Valsalva Maneuver

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design comparing Valsalva maneuver with standard care.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor (dialysis nurse) is blinded to group allocation to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsalva Maneuver Group (Experimental): Patients perform the Valsalva maneuver during AVF cannulation in each dialysis session.
  Interventions: Behavioral: Valsalva Maneuver
- Control Group (No Intervention): Patients receive standard AVF cannulation care without any additional intervention.

INTERVENTIONS:
Behavioral: Valsalva Maneuver — Patients are instructed to perform the Valsalva maneuver by blowing into a 10-cc syringe to generate approximately 20 mmHg pressure for 15-20 seconds before arteriovenous fistula cannulation during each dialysis session.
  Arms: Valsalva Maneuver Group

SUMMARY:
The goal of this clinical trial is to evaluate whether the Valsalva maneuver reduces invasive pain during arteriovenous fistula (AVF) cannulation in adult hemodialysis patients. The main questions it aims to answer are:

Does the Valsalva maneuver effectively reduce pain intensity during AVF cannulation as measured by the Visual Analogue Scale (VAS)?

Is the Valsalva maneuver feasible, acceptable, and satisfactory for patients, and can it be sustainably implemented over multiple sessions?

Researchers will compare patients performing the Valsalva maneuver (intervention group) with those receiving standard care without any intervention (control group) to see if pain scores are significantly lower and whether patients are willing to continue using this technique voluntarily.

Participants will:

Receive training and supervised practice on the Valsalva maneuver before inclusion in the study

Perform the Valsalva maneuver during AVF cannulation in each hemodialysis session for 12 sessions

Complete VAS pain assessments after each session

Complete a patient satisfaction and feasibility form at the end of the study

DETAILED DESCRIPTION:
Arteriovenous fistula (AVF) cannulation is a frequent and essential procedure for patients receiving maintenance hemodialysis, yet it often causes moderate to severe pain and anxiety, which can negatively affect patients' treatment adherence and quality of life. Although pharmacological methods are commonly used to manage cannulation-related pain, they can be costly and have potential side effects. Therefore, there is increasing interest in simple, low-cost, non-pharmacological techniques.

The Valsalva maneuver is a physiological technique that increases intrathoracic pressure through forced exhalation against a closed airway, stimulating the vagus nerve and providing an antinociceptive effect. Previous studies have shown that the Valsalva maneuver reduces pain in various invasive procedures such as intravenous cannulation and spinal puncture; however, evidence for its efficacy during AVF cannulation in hemodialysis patients is limited and methodologically weak.

This randomized controlled, single-blind trial aims to evaluate the effectiveness of the Valsalva maneuver in reducing pain intensity during AVF cannulation among adult hemodialysis patients. The study also investigates the feasibility, sustainability, and patient satisfaction associated with the use of this maneuver.

Patients in the intervention group will receive training on the Valsalva maneuver and perform it during each cannulation session over 12 hemodialysis sessions. Pain intensity will be measured using the Visual Analogue Scale (VAS) immediately after each session. At the end of the study, patient feedback regarding the acceptability and ease of use of the maneuver will be collected through a structured form.

This study is designed to provide high-level evidence supporting a cost-effective, easily applicable, and non-pharmacological approach to pain management during AVF cannulation, potentially contributing to improved patient comfort and adherence to hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receiving hemodialysis treatment via arteriovenous fistula for at least 3 months
* No analgesic medication use within the past 24 hours
* Systolic blood pressure between 90-160 mmHg and diastolic between 60-100 mmHg
* Pain score ≥ 1 on Visual Analogue Scale during AVF cannulation
* Able to perform the Valsalva maneuver (no contraindications)
* No communication barriers or severe psychiatric disorders
* Provided written informed consent

Exclusion Criteria:

* Unable to correctly perform the Valsalva maneuver
* Failed first cannulation attempt
* History of acute myocardial infarction or malignant arrhythmia
* Aneurysm, infection, edema, or scar tissue at AVF site
* Pregnancy
* Voluntary withdrawal from the study at any stage
* Switching dialysis centers or requiring hospitalization during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity During AVF Cannulation Assessed by Visual Analogue Scale (VAS) | Up to 12 hemodialysis sessions (approximately 3 months)
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), a 0-10 scale where 0 means no pain and 10 means the worst possible pain, immediately after each AVF cannulation session.

SECONDARY OUTCOMES:
Patient Satisfaction With the Valsalva Maneuver | At the end of 12 hemodialysis sessions (approximately 3 months)
  Patient satisfaction regarding the feasibility, comfort, and willingness to continue using the Valsalva maneuver will be assessed through a structured satisfaction form at the end of the study period.
Feasibility of Performing the Valsalva Maneuver | Up to 12 hemodialysis sessions (approximately 3 months)
  The feasibility of performing the Valsalva maneuver will be evaluated based on patients' ability to correctly perform the maneuver and their reports of any difficulties during the study period.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request for meta-analysis purposes after publication of the primary results.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of primary results; available for up to 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal and agree to use the data only for meta-analysis or pooled analysis purposes. Requests should be directed to the principal investigator.

REFERENCES:
- [Background] Babamohamadi H, Ameri Z, Asadi I, Asgari MR. Comparison of the Effect of EMLA Cream and the Valsalva Maneuver on Pain Severity during Vascular Needle Insertion in Hemodialysis Patients: A Controlled, Randomized, Clinical Trial. Evid Based Complement Alternat Med. 2022 Aug 31;2022:8383021. doi: 10.1155/2022/8383021. eCollection 2022. PMID 36091600
- [Background] Hosseini SJ, Manzari ZS, Karkhah S, Heydari A. The effects of Valsalva maneuver on pain intensity and hemodynamic status during short peripheral cannula insertion in adults: A systematic review and meta-analysis. J Vasc Access. 2024 Jul;25(4):1051-1062. doi: 10.1177/11297298221145982. Epub 2022 Dec 27. PMID 36573708
- [Result] Alzaatreh MY, Abdalrahim MS. Management Strategies for Pain Associated with Arteriovenous Fistula Cannulation: An Integrative Literature Review. Hemodial Int. 2020 Jan;24(1):3-11. doi: 10.1111/hdi.12803. Epub 2019 Dec 3. PMID 31797508